CLINICAL TRIAL: NCT02255318
Title: Primary Prevention of Infections Related to Chambers Implantable Catheter by a Taurolodine Lock in Patients With Cancer Receiving Parenteral Nutrition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2013-792
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Cancer; Infection
Keywords: Taurolock®; infections related to chambers implantable catheter; patients with cancer receiving parenteral nutrition
MeSH Terms: conditions — Neoplasms; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Taurolock (Experimental): Patients received Taurolock lock for 3 months administration.
  Interventions: Device: Taurolock
- Placebo (Placebo Comparator): Patients received placebo lock (physiological serum) for 3 months administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Device: Taurolock
  Arms: Taurolock
Drug: Placebo
  Arms: Placebo

SUMMARY:
The therapeutic management of patients with cancer often requires the establishment of a chamber implantable catheter. Infections are the main complication of these catheters. These infections may be responsible for a significant impairment of quality of life for patients, and may increase the frequency and duration of hospitalizations. The rate of mortality from these infections is about 17%. The objective of this study is to evaluate the efficacy of a 1.35% taurolidine lock / 4% citrate (TauroLock®) in the primary prevention of infections related to chambers implantable catheter (IRCIC) in cancer patients receiving parenteral nutrition.

This is a, randomized, double-blind clinical trial comparing the incidence of IRCIC in patients receiving Taurolidine lock or concession the usual procedure of rinsing with saline (placebo) (pulsed rinsing with 20 mL of serum physiological and clamping catheter positive pressure). The lock will be instilled after the end of the session IV treatment (chemotherapy, parenteral nutrition, transfusion) before closing the catheter. The primary endpoint will be the rate IRCIC in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over
* Patients with solid cancer
* Patients with implantable catheter
* Patients receiving parenteral nutrition
* Patient affiliated to a social security scheme or beneficiary of such a regime

Exclusion Criteria:

* Patients refusing to participate in the protocol
* Patients already receiving preventive lock of IRCIC
* Known citrate or (cyclo) allergy -taurolidine
* Patients taking other drugs with known contraindications against the citrate or cyclotaurolidine.
* Participation in another protocol for the prevention of infections associated with central venous catheters
* Patients who did not sign the consent
* Patient with a status of socio-legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of infections related to chamber implantable catheters (IRCIC) in patients who received Taurolock® versus those who received the usual procedure of saline flush. | The incidence will be assessed between the inclusion and 3 months after the beginning of the study.
  Definition of IRCIC This definition of infections related to chamber implantable catheters will be used for all patients. It is based on the identification of the same germ blood cultures of peripheral vein and those of the central venous line with a differential time greater than 120 minutes growth.

SECONDARY OUTCOMES:
Delay onset of IRCIC | between the inclusion and 3 months after the beginning of the study
Duration of hospitalizations for IRCIC. | between the inclusion and 3 months after the beginning of the study

CONTACTS AND LOCATIONS:
Overall Officials: Cécile CHAMBRIER, PH, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Hôpital Edouard Herriot, France, Lyon
  - Hôpital de la Croix Rousse, France
  - Groupement Hospitalier Lyon Sud, Pierre-Bénite